CLINICAL TRIAL: NCT01596985
Title: Prospective, Monocentric Study Comparing Cystectomy to PlasmaJet Ablation in the Surgical Management of Ovarian Endometriomas
Brief Title: Ovarian Endometrioma Ablation Using Plasma Energy Versus Cystectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Plasma Surgical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.S.PJ.6.10.GYN
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Ovarian Endometrioma
Keywords: Endometrioma; Endometriosis; Cystectomy; Ablation; Plasma energy
MeSH Terms: conditions — Endometriosis | interventions — Cystectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ablation using the PlasmaJet system (Experimental): Origin of cyst invagination is identified after lysis of adhesions between ovary and adjacent broad ligament, leading to characteristic "chocolate fluid" evacuation. Surgeon then attempts to turn cyst completely inside out via original invagination site of diameter averaging 1 to 2cm. Ablation of cyst's inner surface is performed using the PlasmaJet system in coagulation mode set at 40, at distance averaging 5mm from tip of handpiece, and with exposure time limited to 1 to 2s on each site. Care is taken not to leave any untreated sites and to ablate the edges of the invagination site and corresponding peritoneal implants on adjacent broad ligament. When cyst reversion is not feasible, surgeon progressively exposes cyst interior to guide plasma beam at an angle perpendicular to the inner surface.
  Interventions: Procedure: Ablation using the PlasmaJet system
- Cystectomy (Active Comparator): Surgical excision of an ovarian endometrioma by cystectomy involves three distinct areas, each requiring a different excision procedure. Area A from where cyst invagination originates, measures 1 cm² on average and is revealed by lysing adhesions between the ovary and the adjacent broad ligament, leading to the characteristic "chocolate fluid" evacuation. The excision by scissors of area A allows the surgeon to identify a cleavage plane close to the cyst wall, which can be followed without significant bleeding (area B). Should adhesions appear in the cleavage plane, they are coagulated and cut, so as not to strip the ovarian cortex. Close to the ovarian hilus, for complete cyst removal, adhesions require coagulation using bipolar current and section by scissors (area C).
  Interventions: Procedure: Cystectomy

INTERVENTIONS:
Procedure: Ablation using the PlasmaJet system — Ablation of the inner surface of the cyst is then performed using the PlasmaJet system in coagulation mode set at 40, at a distance averaging 5 mm from the tip of the handpiece, and with an exposure time limited to 1 to 2 seconds on each site. Care is taken not to leave any untreated sites and to ablate the edges of the invagination site and the corresponding peritoneal implants on the adjacent broad ligament.
  Other Names: Ovarian cyst ablation; Ablation by plasma energy
  Arms: Ablation using the PlasmaJet system
Procedure: Cystectomy — Surgical excision of an ovarian endometrioma by cystectomy involves three distinct areas, each requiring a different excision procedure. Area A from where cyst invagination originates, measures 1 cm² on average and is revealed by lysing adhesions between the ovary and the adjacent broad ligament, leading to the characteristic "chocolate fluid" evacuation. The excision by scissors of area A allows the surgeon to identify a cleavage plane close to the cyst wall, which can be followed without significant bleeding (area B). Should adhesions appear in the cleavage plane, they are coagulated and cut, so as not to strip the ovarian cortex. Close to the ovarian hilus, for complete cyst removal, adhesions require coagulation using bipolar current and section by scissors (area C).
  Other Names: Cyst excision; Ovarian stripping
  Arms: Cystectomy

SUMMARY:
Objective: To compare loss of ovarian parenchyma following ovarian endometrioma ablation using the PlasmaJet system versus cystectomy, using postoperative examination by 3D ultrasound.

Design: Prospective comparative study. Setting: Two experienced surgeons practicing in two University tertiary referral centers.

Patients: Fifty women with no previous history of ovarian surgery managed for unilateral ovarian endometrioma > 30 mm in diameter.

Interventions: Endometrioma ablation by plasma energy using the PlasmaJet system and ovarian tissue sparing cystectomy.

Main Outcome Measures: 3D ultrasound assessment of postoperative reduction in ovarian volume and antral follicle count (AFC) .

DETAILED DESCRIPTION:
The management of ovarian endometriomas in women wishing to conceive remains challenging. Recent data suggest that excising endometriomas by ovarian tissue sparing cystectomy does not avoid inadvertent removal of ovarian parenchyma surrounding the cyst, particularly in enlarged cysts. Although several authors question whether the ovarian parenchyma immediately surrounding the cyst may still be functional, there is little doubt that postoperative fertility could be significantly impaired by loss of ovarian cortex and provokes the question as to whether pregnancy should be initiated before performing a cystectomy, whenever this scenario is possible. However ovarian surgery cannot always be delayed to the postpartum period, numerous women require endometrioma management while not seeking an immediate pregnancy and still wish to conserve their procreative capabilities.

After a period of some years during which cystectomy appeared to be the best surgical technique in the treatment of ovarian endometriomas in women wishing to become pregnant, recent data have suggested that ablation of the inner layer of the endometrioma may be a valuable alternative technique, as long as the energy employed avoids thermal diffusion to surrounding ovarian tissue. The Department of Gynecology at the University Hospital in Rouen, France have introduced ablation by plasma energy using the PlasmaJet system (Plasma Surgical Ltd, Abingdon, UK) and have already been able to report encouraging results based on non comparative pilot studies and on retrospective "before and after" comparative study.

The aim of the study is to prospectively compare loss of ovarian parenchyma and decrease in antral follicle count (AFC) following ovarian endometrioma ablation using plasma energy versus cystectomy, when performed by only two expert surgeons. Postoperative examination is carried out by 3D ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years;
* Surgery required by pelvic pain or infertility related to endometriosis;
* Clinical and imaging data proving unilateral ovarian endometrioma which diameter exceeds 30 mm.

Exclusion Criteria:

* Previous surgery on ovaries or IVF procedures;
* Bilateral endometriomas;
* Pregnancy
* Woman not French speaker.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Loss of ovarian volume | 3 months postoperatively
  Evaluation of ovarian volumes of both the operated and the contralateral healthy ovary using a tridimensional ultrasound by vaginal route. The volume of each ovary expressed in cm³ was estimated using the formula D1 x D2 x D3 x π / 6. The Mann and Whitney test is performed to compare measurements made on the operated ovaries vs. those made on the contralateral ovaries.

SECONDARY OUTCOMES:
Decrease in ovarian antral follicles count (AFC) | 3 months postoperatively
  Evaluation of antral follicle counts in both the operated and the contralateral, healthy ovary, using tridimensional ultrasound. The Mann and Whitney test is performed to compare the decrease in AFC depending on surgical procedure.
Antimullerian Hormone level (AMH) | 3 months postoperatively
  AMH level are measured before and 3 months after the surgery to evaluate the decrease in AMH level depending on surgical technique.

CONTACTS AND LOCATIONS:
Overall Officials: Horace Roman, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - University Hospital, Clermont-Ferrand, Auvergne
  - University Hospital, Rouen, Seine-Maritime

REFERENCES:
- [Derived] Roman H, Bubenheim M, Auber M, Marpeau L, Puscasiu L. Antimullerian hormone level and endometrioma ablation using plasma energy. JSLS. 2014 Jul-Sep;18(3):e2014.00002. doi: 10.4293/JSLS.2014.00002. PMID 25392649